CLINICAL TRIAL: NCT01461564
Title: Randomized Clinical Trial to Compare Air Versus Carbon Dioxide in Screening Unsedated Colonoscopy.
Brief Title: Carbon Dioxide During Screening Unsedated Colonoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Radoslaw Pach, Assisstant Professor, Jagiellonian University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: Cracow CO2 Trial
Record Dates: First submitted 2011-10-26; First posted 2011-10-28 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-06

CONDITIONS: Polyps
Keywords: screening; colonoscopy; carbon dioxide; air; pain score; complications
MeSH Terms: conditions — Polyps | interventions — Colonoscopy; Endoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carbon dioxide (Experimental): Patients insufflated with carbon dioxide during screening colonoscopy
  Interventions: Procedure: Colonoscopy
- Air (Active Comparator): Patients insufflated with air during screening colonoscopy
  Interventions: Procedure: Colonoscopy

INTERVENTIONS:
Procedure: Colonoscopy — Screening colonoscopy
  Other Names: Endoscopy; Flexible endoscopy

SUMMARY:
Colonoscopy is currently most effective procedure used for detecting colon cancer especially in the early stages. Screening colonoscopies are performed in the symptom-free patients at risk of familial colon cancer. During colonoscopy air commonly used to insufflate the bowel may be retained after the procedure causing pain and discomfort to the patients. One of the methods used to reduce pain and discomfort is insufflation of carbon dioxide (CO2) instead of air during colonoscopy.

Aim of the study is evaluation of the use of carbon dioxide insufflation during colonoscopy.

DETAILED DESCRIPTION:
The study was conducted in 200 consecutive patients undergoing screening colonoscopies for the detection of early colon cancer. The examinations were performed with Olympus 165 colonoscopes by seven experienced endoscopists, each of whom performed alone about over 2000 colonoscopies. The patients were randomly assigned to Group I and II with either air or carbon dioxide insufflation. Both study groups were matched by sex, age, duration of the procedure, and BMI. The authors compared for the duration of the procedure, coecal intubation time, complication rate, pulse rates immediately after the procedure, 15 minutes after, and subjective pain evaluation on a Visual Analogue Scale.

ELIGIBILITY:
Inclusion Criteria:

* age 50 yo and more
* no previous large bowel operations
* no previous colonoscopy
* informed consent

Exclusion Criteria:

* previous colonoscopy
* previous large bowel operations/ polypectomies

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
duration of procedure | 1 hour
  Time from introduction of a colonoscope to removal of the colonoscope.

SECONDARY OUTCOMES:
coecal intubation time | 1 hour
  Time from introduction of a colonoscope to intubation of the coecumo
pain immediately after the procedure | 1 min
  Pain assessed by VAS scale immediately after colonoscopy
pain 15 minutes after colonoscopy | 15 min
  Pain assessed by VAS scale 15 minutes after colonoscopy
complication rate | 24 hours
  any compication of screening colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Miroslaw Szura, MD PhD, Study Director — I Dept of General, Oncological and GI Surgery Jagiellonian University; Radoslaw Pach, MD PhD, Principal Investigator — I Dept of General, Oncological and GI Surgery Jagiellonian University; Andrzej Matyja, MD PhD, Study Chair — I Dept of General, Oncological and GI Surgery Jagiellonian University
Locations (1):
- 1st Department of General, Oncological and Gastrointestinal Surgery, Jagiellonian University, Krakow, Malopolska, Poland

REFERENCES:
- [Result] Szura M, Pach R, Matyja A, Kulig J. Carbon dioxide insufflation during screening unsedated colonoscopy: a randomised clinical trial. Eur J Cancer Prev. 2015 Jan;24(1):37-43. doi: 10.1097/CEJ.0000000000000047. PMID 24915135